CLINICAL TRIAL: NCT00169494
Title: Immunogenicity: 3 Consecutive Lots of GSK Biologicals' HPV-16/18 Vaccine Administered Intramuscularly at 0,1,6 Month Schedule in Healthy Females Aged 10-25 Years and Demonstrate Non-inferiority of Candidate HPV Vaccine Manufactured by Modified Production Process
Brief Title: Human Papilloma Virus Vaccine Consistency and Non-inferiority Trial in Young Adult Women With GSK Bio HPV-16/18
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: 580299/012
Record Dates: First submitted 2005-09-12; First posted 2005-09-15 (Estimated); Last update posted 2016-09-12 (Estimated); Status verified 2016-09

CONDITIONS: Infections, Papillomavirus
MeSH Terms: conditions — Papillomavirus Infections

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor

INTERVENTIONS:
Biological: HPV-16/18 L1/AS04

SUMMARY:
Human Papilloma virus (HPV) are viruses that cause a common infection of the skin and genitals in men and women. Several types of HPV infection are transmitted by sexual activity and, in women, can infect the cervix (part of the uterus or womb). This infection often goes away by itself, but if it does not go away (this is called persistent infection), it can lead in women over a long period of time to cancer of the cervix. If a woman is not infected by HPV, it is very unlikely that she will get cervical cancer. This study will evaluate the consistency of consecutive vaccine lots and the non-inferiority of modified manufacturing processes of GSK Biologicals HPV-16/18 vaccine and the vaccine safety, over 12 months, in young adolescents and women of 10-25 years of age at study start. Approximately 750 study subjects will receive different lots of the HPV vaccine administered intramuscularly according to a 0-1-6 month schedule.

ELIGIBILITY:
Inclusion Criteria:

* A woman between, and including, 10 and 25 years of age at the time of the first vaccination.
* Written informed consent from the subject prior to enrolment.
* Subject must be free of obvious health problems.
* Subject must have negative urine pregnancy test.

Exclusion Criteria:

* Pregnant or breastfeeding.
* Known acute or chronic, clinically significant pulmonary, cardiovascular, neurologic, hepatic or renal functional abnormality.
* History of chronic condition(s) requiring treatment such as cancer, chronic hepatitis or kidney disease(s), diabetes, or autoimmune disease.
* Previous vaccination against human papillomavirus (HPV).

Ages: 10 Years to 25 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 770 (Actual)
Dates: Start 2004-09; Primary Completion 2005-07 (Actual); Study Completion 2005-07 (Actual)

PRIMARY OUTCOMES:
Demonstration of lot-to-lot consistency in terms of immunogenicity of 3 lots of HPV-16/18 vaccine.
Demonstration of non-inferiority in terms of immunogenicity of the HPV vaccine produced with a revised manufacturing process compared to the HPV vaccine produced with a previous manufacturing process

SECONDARY OUTCOMES:
Safety of HPV vaccine in entire study period. Immunogenicity bridge between pre-adolescent and adolescent population.

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (14):
- Denmark (2):
  - GSK Investigational Site, Koebenhavn NV
  - GSK Investigational Site, Odense C
- Estonia (2):
  - GSK Investigational Site, Tallinn
  - GSK Investigational Site, Tartu
- Finland (2):
  - GSK Investigational Site, Seinäjoki
  - GSK Investigational Site, Tampere
- Greece (3):
  - GSK Investigational Site, Athens
  - GSK Investigational Site, Heraklion, Crete
  - GSK Investigational Site, Thessaloniki
- GSK Investigational Site, Rotterdam, Netherlands
- Russia (4):
  - GSK Investigational Site, Kazan'
  - GSK Investigational Site, Moscow
  - GSK Investigational Site, Smolensk
  - GSK Investigational Site, Volgograd

IPD SHARING:
Plan to Share IPD: Yes
Patient-level data for this study will be made available through www.clinicalstudydatarequest.com following the timelines and process described on this site.

REFERENCES:
- [Derived] Lehtinen M, Lagheden C, Luostarinen T, Eriksson T, Apter D, Bly A, Gray P, Harjula K, Heikkila K, Hokkanen M, Karttunen H, Kuortti M, Nieminen P, Nummela M, Paavonen J, Palmroth J, Petaja T, Pukkala E, Soderlund-Strand A, Veivo U, Dillner J. Human papillomavirus vaccine efficacy against invasive, HPV-positive cancers: population-based follow-up of a cluster-randomised trial. BMJ Open. 2021 Dec 30;11(12):e050669. doi: 10.1136/bmjopen-2021-050669. PMID 35149535
- See also: Month 18 FU — http://clinicaltrials.gov/ct/show/NCT00337818?order=1
- See also: Month 24 FU — http://clinicaltrials.gov/ct/show/NCT00337818?order=1
- See also: Month 36 FU — http://clinicaltrials.gov/ct/show/NCT00337818?order=1
- See also: Month 48 FU — http://clinicaltrials.gov/ct/show/NCT00337818?order=1
- Available data/document: Informed Consent Form: 580299/012 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Dataset Specification: 580299/012 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Annotated Case Report Form: 580299/012 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Clinical Study Report: 580299/012 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Statistical Analysis Plan: 580299/012 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Study Protocol: 580299/012 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Individual Participant Data Set: 580299/012 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register. The results of this study 580299/012 are summarised with studies 107476 (M18), 107477 (M24), and 107479 (M36) on the GSK Clinical Study Register.